CLINICAL TRIAL: NCT03420638
Title: Randomized Clinical Trial Examining Use of Adjunct EXPAREL for Post-tonsillectomy Pain Management in Adults
Brief Title: EXPAREL Post-tonsillectomy Clinical Trial
Acronym: EXPCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul Hoff (Other)
Collaborators: St. Joseph Mercy Ann Arbor (Unknown)
Responsible Party: Sponsor-Investigator, Paul Hoff, Principal Investigator, Trinity Health Michigan
Organization: Trinity Health Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSR-17-1714
Record Dates: First submitted 2017-10-17; First posted 2018-02-05 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Tonsillectomy
Keywords: Adults; Pain
MeSH Terms: conditions — Pain | interventions — Standard of Care; Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Using sealed envelope assignment, the participant will be placed in study Arm 1 or 2. The PI will not be masked because the PI will administer the adjunct treatment or the standard of care only. The outcome assessor will be masked to study group assignment for gathering data from trial participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunct Exparel (Experimental): After removal of the tonsils and before extubation, the principal investigator will infiltrate 0.5 mL of the standard of care medication-bupivacaine HCl 0.25% (2.5 mg/mL) with epinephrine (5 mcg/mL) i.m.-into the upper and lower poles of the anterior and posterior tonsillar pillars on the right and left side of the oropharynx for a volume of 2 mL of bupivacaine HCl on each side. Following the standard medication, the principal investigator will infiltrate 0.5 mL of adjunct Exparel (bupivacaine liposome suspension 1.3% [13.3 mg/mL], i.m.) into the upper and lower poles of the anterior and posterior tonsillar pillars on the right and left side of the oropharynx for a volume of 2 mL of bupivacaine liposome injectable suspension on each side.
  Interventions: Drug: Adjunct Exparel (bupivacaine liposome suspension 1.3%); Other: Standard Care
- Standard Care (Other): After removal of the tonsils and before extubation, the principal investigator will infiltrate 0.5 mL of the standard of care medication-bupivacaine HCl 0.25% (2.5 mg/ mL) with epinephrine (5 mcg/mL) i.m.-into the upper and lower poles of the anterior and posterior tonsillar pillars on the right and left side of the oropharynx for a volume of 2 mL of bupivacaine HCl on each side.
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: Adjunct Exparel (bupivacaine liposome suspension 1.3%) — After removal of the tonsils and before extubation, the principal investigator will infiltrate 0.5 mL of the standard of care medication-bupivacaine HCl 0.25% (2.5 mg/mL) with epinephrine (5 mcg/mL) i.m.-into the upper and lower poles of the anterior and posterior tonsillar pillars on the right and left side of the oropharynx for a volume of 2 mL of bupivacaine HCl on each side. Following the standard medication, the principal investigator will infiltrate 0.5 mL of adjunct Exparel (bupivacaine liposome suspension 1.3% [13.3 mg/mL] i.m.) into the upper and lower poles of the anterior and posterior tonsillar pillars on the right and left side of the oropharynx for a volume of 2 mL of bupivacaine liposome injectable suspension 1.3% (13.3 mg/mL) on each side.
  Other Names: Bupivacaine liposome suspension 1.3%
  Arms: Adjunct Exparel
Other: Standard Care — After removal of the tonsils and before extubation, the principal investigator will infiltrate 0.5 mL of the standard of care medication-bupivacaine HCl 0.25% (2.5 mg/ mL) with epinephrine (5 mcg/mL) i.m.-into the upper and lower poles of the anterior and posterior tonsillar pillars on the right and left side of the oropharynx for a volume of 2 mL of bupivacaine HCl on each side.
  Other Names: Bupivacaine HCl with epinephrine

SUMMARY:
Tonsillectomy is one of the most commonly performed surgical procedures in the United States. The primary indications for tonsillectomy in the adult population include recurrent pharyngitis, chronic tonsillitis, and obstructive pathology. Tonsillectomy is often associated with severe postoperative pain, which can result in prolonged poor oral intake, dehydration, and the need for high dose narcotics. In severely dehydrated patients, epithelial shedding and necrosis of soft tissues at the surgical site can lead to postoperative complications such as bleeding, delayed healing, and severe pain. The goal for this study is to explore the use of a long acting local anesthetic bupivacaine liposome injectable suspension (Exparel) to manage pain experienced by adult patients after tonsillectomy

DETAILED DESCRIPTION:
The proposed investigation will examine whether Exparel (bupivacaine liposome injectable suspension 1.3%-13.3 mg/mL) when used as a post-excision adjunct to the standard of care bupivacaine HCl 0.25% (2.5 mg/mL) with Epinephrine (5mcg/mL), will decrease the patient's post-tonsillectomy experience of pain intensity, especially for the first three days after surgery, and correspondingly reduce the requirement for pain medications and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo bilateral palatine tonsillectomy as the only procedure
2. Adults age 18 years and older.

Exclusion Criteria:

1. Severe systemic disease that is clinically significant in the judgement of the investigator.
2. Coagulation disorder that is clinically significant in the judgement of the investigator.
3. Current or previous history of analgesic dependence
4. Allergy to any of the drugs used in the study (bupivacaine)
5. Women known to be pregnant, planning to become pregnant, or lactating
6. Hearing impairment that is clinically significant in the judgement of the investigator.
7. Cardiovascular disease that is clinically significant in the judgement of the investigator.
8. Impaired liver function that is clinically significant in the judgement of the investigator.
9. Impaired renal function that is clinically significant in the judgement of the investigator.
10. Unable to provide consent.
11. Additional surgical procedures planned concurrently with palatine tonsillectomy.
12. Planned use of topical or injected anesthetics other than those administered by the study within the two week follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain rating between post anesthesia care unit (PACU) baseline and designated post-operative days | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported average and maximum pain rating over a 24-hour period using the St. Joseph Mercy Ann Arbor (SJMAA) standard visual analog 11 point pain rating scale. The minimum value of 0 indicates no pain and the maximum value of 10 indicates the worst possible pain. A higher value represent greater pain and a worse outcome. The baseline pain rating is the maximum rating from PACU on the day of surgery. Day-1 begins at 12:00 AM (after midnight) day of surgery and extends through 11:59 PM. Each following designated day will begin at 12:00 AM and extend through 11:59 PM.

SECONDARY OUTCOMES:
Change in total amount of prescribed narcotic pain medication taken between Day-1 and designated post-operative days | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported amount of prescribed narcotic pain medication in mg. taken during a 24-hour period. Higher values represent greater amounts of narcotic pain medication consumed and a worse outcome. Day-1 begins at 12:00 AM (midnight after the day of surgery and extends through 11:59 PM. Day-2 and each following designated day will begin at 12:00 AM and will extend through 11:59 PM.
Change in the total amount of over the counter pain medication taken between Day-1 and designated post-operative days | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported amount of over the counter pain medication taken in mg during a 24-hour period. Higher values represent greater amounts of over the counter pain medication consumed and a worse outcome. Day-1 begins at 12:00 AM (after midnight) day of surgery and will extend through 11:59 PM. Day-2 and each following designated day will begin at 12:00 AM and will extend through 11:59 PM.

OTHER OUTCOMES:
Change in the amount of fluid intake consumed between Day-1 and designated post-operative days | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported amount of fluid intake in ounces during a 24-hour period. Lower values represent less fluid intake and a worse outcome.
Time to change in food intake | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported time in days to change in food intake from liquids to other thicker foods such as smoothies, cream soups, puddings, etc., and to solid food such as eggs, mashed vegetables, soft pasta, etc. A longer duration until a change in food intake represents a worse outcome.
Time to first physical activity outside of the home | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported day of first physical activity outside of the home, such as running an errand. A longer duration until physical activity outside of the home represents a worse outcome.
Adverse Event | Post-tonsillectomy Days 1, 2, 3, 5, and 10
  Patient reported adverse event such as bleeding, Emergency Department visit, return to surgery, allergic reaction, side effects of medication, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - St. Joseph Mercy Ann Arbor, Ann Arbor, Michigan
  - Michigan Otolaryngology Surgery Associates, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2. Marcaine™ [package insert]. Hospira, Inc., Lake Forest, IL; October 2011. https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/022046s004lbl.pdf. Accessed June 12, 2017.
- [Background] Bulbake U, Doppalapudi S, Kommineni N, Khan W. Liposomal Formulations in Clinical Use: An Updated Review. Pharmaceutics. 2017 Mar 27;9(2):12. doi: 10.3390/pharmaceutics9020012. PMID 28346375
- [Result] 1. Exparel® [package insert]. Pacira Pharmaceuticals, Inc., San Diego, CA; 2015. https://www.exparel.com/sites/default/files/EXPAREL_Prescribing_Information.pdf. Accessed June 12, 2017.
- [Result] Cullen KA, Hall MJ, Golosinskiy A. Ambulatory surgery in the United States, 2006. Natl Health Stat Report. 2009 Jan 28;(11):1-25. PMID 19294964
- [Result] Grainger J, Saravanappa N. Local anaesthetic for post-tonsillectomy pain: a systematic review and meta-analysis. Clin Otolaryngol. 2008 Oct;33(5):411-9. doi: 10.1111/j.1749-4486.2008.01815.x. PMID 18983373
- [Result] Bhattacharyya N, Kepnes LJ. Revisits and postoperative hemorrhage after adult tonsillectomy. Laryngoscope. 2014 Jul;124(7):1554-6. doi: 10.1002/lary.24541. Epub 2014 Jan 3. PMID 24281921
- [Result] Stelter K, Hiller J, Hempel JM, Berghaus A, Hagedorn H, Andratschke M, Canis M. Comparison of two different local anaesthetic infiltrations for postoperative pain relief in tonsillectomy: a prospective, randomised, double blind, clinical trial. Eur Arch Otorhinolaryngol. 2010 Jul;267(7):1129-34. doi: 10.1007/s00405-009-1200-8. Epub 2010 Jan 13. PMID 20069307
- [Result] Arikan OK, Ozcan S, Kazkayasi M, Akpinar S, Koc C. Preincisional infiltration of tonsils with ropivacaine in post-tonsillectomy pain relief: double-blind, randomized, placebo-controlled intraindividual study. J Otolaryngol. 2006 Jun;35(3):167-72. PMID 16929992
- [Result] Diakos EA, Gallos ID, El-Shunnar S, Clarke M, Kazi R, Mehanna H. Dexamethasone reduces pain, vomiting and overall complications following tonsillectomy in adults: a systematic review and meta-analysis of randomised controlled trials. Clin Otolaryngol. 2011 Dec;36(6):531-42. doi: 10.1111/j.1749-4486.2011.02373.x. PMID 21812940
- [Result] 10. Tamm-Daniels, Inge. Liposomal Bupivacaine: What Is All The Fuss? University of Wisconsin School of Medicine and Public Health Madison, 5 Nov 2014-video Department of Anesthesiology grand Rounds https://videos.med.wisc.edu/videos/56752. Accessed July 10, 2017.
- [Result] Tong YC, Kaye AD, Urman RD. Liposomal bupivacaine and clinical outcomes. Best Pract Res Clin Anaesthesiol. 2014 Mar;28(1):15-27. doi: 10.1016/j.bpa.2014.02.001. Epub 2014 Mar 15. PMID 24815964